CLINICAL TRIAL: NCT04965259
Title: Early Detection of Hepatocellular Carcinoma (HCC): miRNA, Microbiome and Imaging Biomarkers in the Evolution of Chronic Liver Disease in a High-risk Prospective Cohort (ELEGANCE)
Brief Title: Early Detection of Hepatocellular Carcinoma in a High-risk Prospective Cohort (ELEGANCE)
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore Phenome Centre (Unknown); Nanyang Technological University (Other); MiRXES Pte Ltd (Industry); Perspectum Asia Pte Ltd (Unknown); Asian Microbiome Library Pte Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: AHCC10 ELEGANCE
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Liver Diseases
Keywords: Hepatocellular Carcinoma(HCC); Surveillance; Patients-at-risk; miRNA; Precision medicine; Gut microbiota; Metabolites; Microbiome biomarkers; Circulating biomarkers; MRI
MeSH Terms: conditions — Liver Diseases; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloods shall be used for relevant laboratory assessments. Blood, urine and stool samples shall be used for miRNA, microbiome and metabolome profiling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) is the 7th most common cause of cancer death globally but only 20% are diagnosed in its early stages where cure is possible. Current standard-of-care surveillance of patients at high risk of developing HCC with 6-monthly serum alpha-fetoprotein (AFP) and ultrasound imaging (US) has a sensitivity of approximately 63% for detecting early HCC. There is an urgent need for a more efficacious and convenient modality of surveillance of high-risk patients to diagnose HCC at an early stage.

This prospective study aims to address this unmet clinical need by validating a panel of circulating miRNA biomarkers to develop an in-vitro diagnostic (IVD) kit for the detection of early HCC in a cohort of high-risk patients.

Additionally, this study also aims to develop a multi-parametric MRI-based AI algorithm to quantify individual risks of developing HCC and to predict the progression of chronic liver disease in this cohort to enable targeted surveillance. Lastly, by identifying changes in the microbiome and metabolites as HCC develops in this cohort enables the establishment of actionable biomarkers that can prevent and predict the development of HCC.

DETAILED DESCRIPTION:
Eligible patients will receive 6-monthly standard-of-care surveillance (US, serum AFP and liver function test) for HCC until end of study or up to a maximum of 7 assessments (1 baseline and 6 follow-up assessments). There will be an option for patients to continue to receive standard-of-care surveillance for HCC until end of study or up to 6 additional assessments (Visits 8-13), whichever occurs first.

Patients with elevated AFP or abnormalities detected on US will be investigated with multi-phasic CT scan or MRI to confirm or refute the diagnosis of HCC. Additionally, patients shall be scheduled for sequential bio-samples collection (blood, urine and stool) and blood tests (Hba1c and Lipid Panel) during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 50 to 90 years of age at the time of signing the informed consent form, except for patients recruited under the cirrhotic group, patients of 40 to 90 years of age can be included.
* Patient has serum alpha-fetoprotein (AFP) within normal range of the investigating laboratory in the past 3 months. For patients with AFP level out of the normal range of the investigating laboratory and up to 15.0ug/L, patient will be eligible if patient has a CT/MRI scan that exclude HCC in the past 3 months.
* Patient has ultrasound hepatobiliary system (US HBS) that does not show lesion suspicious for HCC or, CT / MRI scan that exclude HCC, in the past 3 months
* Patient is estimated to survive more than 3 years
* Patient with any of the following chronic liver disease:

  1. liver cirrhosis of any etiology, identified by elastography (liver stiffness > 13 kPa), US, CT, MRI or liver biopsy, Child-Pugh class A and B
  2. non-cirrhotic chronic viral hepatitis (B or C) or both
  3. non-alcoholic fatty liver disease (NAFLD)
  4. non-alcoholic steatohepatitis (NASH)
* Patient is able to comply with scheduled visits, assessments and other study procedures
* Patient is willing to provide informed consent before enrolment in the study

Exclusion Criteria:

* Patient with confirmed diagnosis of HCC by the American Association for the Study of the Liver Disease (AASLD) imaging criteria or histology / cytology within the last 5 years
* Patient with Child-Pugh C cirrhosis at time of enrolment (based on the judgement of the Investigator)
* Patient with active hepatic encephalopathy at time of enrolment
* Patient is known to be positive for the Human Immunodeficiency Virus (HIV)
* Patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures
* Patient is unable to provide informed consent or refuse blood taking
* Patient has any other condition which, in the opinion of the Investigators, would make the patient unsuitable for enrolment or could interfere with completion of the study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high-risk of developing HCC forming a cohort of patients with cirrhosis from any etiology, chronic hepatitis B without significant cirrhosis, chronic hepatitis C without significant cirrhosis and NAFLD/NASH without significant cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 2002 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Changes in the profile of circulating micro-RNA biomarkers as high-risk patients develop HCC | Baseline and every 6 months thereafter, and at HCC diagnosis every 6 months thereafter up to 70 months.
  Changes in the profile of circulating micro-RNA biomarkers as high-risk patients develop HCC
value of cT1, PDFF and T2* levels to predict individual's risk of developing and progression of HCC. | Baseline and upon elevated AFP or US which is suggestive of HCC, up to 70 months.
  value of cT1, PDFF and T2* levels to predict individual's risk of developing and progression of HCC.
Changes in the profile of gut microbiota as high-risk patients develop HCC. | Baseline and every 6 months thereafter, up to 70 months
  Changes in the profile of gut microbiota as high-risk patients develop HCC.
Changes in the profile of metabolome in urine and plasma as high-risk patients develop HCC. | Baseline and every 6 months thereafter, up to 70 months.
  Changes in the profile of metabolome in urine and plasma as high-risk patients develop HCC.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (14):
- Singapore (14):
  - National University Hospital, Singapore
  - SingHealth Polyclinics - Bukit Merah, Singapore
  - National Cancer Center Singapore, Singapore
  - SingHealth Polyclinics - Outram, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - SingHealth Polyclinics - Marine Parade, Singapore
  - SingHealth Polyclinics - Bedok, Singapore
  - SingHealth Polyclinics - Pasir Ris, Singapore
  - SingHealth Polyclinics - Tampines, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - SingHealth Polyclinics - Sengkang, Singapore
  - SingHealth Polyclinics - Punggol, Singapore

IPD SHARING:
Plan to Share IPD: Undecided